CLINICAL TRIAL: NCT01445262
Title: Drug Use Investigation for XYZAL
Brief Title: Drug Use Investigation for XYZAL®
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115066
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
MeSH Terms: conditions — Rhinitis | interventions — levocetirizine

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed levocetirizine tablets: Subjects prescribed levocetirizine tablets for treatment of allergic rhinitis, urticaria, eczema, dermatitis, skin irritation, prurigo or pruritus cutaneous
  Interventions: Drug: Levocetirizine

INTERVENTIONS:
Drug: Levocetirizine

SUMMARY:
This post-marketing surveillance study (PMS) is conducted to collect safety and efficacy data among subjects with allergic rhinitis, urticaria, eczema, dermatitis, skin irritation, prurigo or pruritus cutaneous who have never been treated with levocetirizine tablets before.

ELIGIBILITY:
Inclusion Criteria:

* Must be the first time for taking levocetirizine tablet

Exclusion Criteria:

* As this is PMS study, there are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese male and female subjects without age restriction who were considered appropriate to prescribe levocetirizine tablet according to the prescribing information were eligible for this surveillance study.
Sampling Method: Probability Sample
Enrollment: 10728 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects treated with levocetirizine tablets | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline